CLINICAL TRIAL: NCT06418009
Title: Determination of the Effect of Cold Needle Application on Invasive Pain Associated With Fistula Cannulation
Brief Title: Determination of the Effect of Cold Needle on Invasive Pain Cannulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Associate Professor, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2024/50
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hemodialysis Complication; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Pain assessment will be made by a nurse independent of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Not cold needle application (No Intervention): Fistül girişimi için kullanılan iğne kendi torbasında durdurulur ve hastalığın takılacağı zaman Resmi tarafından deponun içinden çıkarılarak kullanılacaktır
- Cold needle application (Experimental): Before use, the needle will be removed from the refrigerator and kept on the nurse's table. When the temperature of the needle reaches 0-2 °C, the patient will be cannulated.
  Interventions: Procedure: Cold needle application

INTERVENTIONS:
Procedure: Cold needle application — Before use, the needle will be removed from the refrigerator and kept on the nurse's table. When the temperature of the needle reaches 0-2 °C, the patient will be cannulated.
  Arms: Cold needle application

SUMMARY:
In studies evaluating the methods used to reduce invasive pain associated with cannulation, it is seen that pharmacological and non-pharmacological methods are used. Pharmacological treatment is considered risky as it may cause drug addiction in the patient and may cause side effects and complications. On the other hand, the use of non-pharmacological methods is preferred because they are cheaper and cause fewer side effects and complications.

DETAILED DESCRIPTION:
Cold application, one of the non-pharmacological methods used, is effective in relieving pain by slowing down or blocking the conduction of peripheral nerves. Apart from this effect, it stimulates touch receptors by activating the Door-Control mechanism; It increases the release of endogenous opioids and stops pain by ensuring the nerve impulses caused by cold are transmitted to Delta fibers. Although studies conducted on hemodialysis patients have shown that cold application is effective in reducing pain; Due to the small number of sample groups and deficiencies in the methodology, it was suggested that further studies be conducted. In these studies, cold application; It was applied to the area one cm above the fistula or between the thumb and index finger of the opposite arm, using an ice pack and an ice-filled glove for 2-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years and older
* had been treated with HD for at least 3 months, thrice a week, and for 4 hours per session
* did not have a psychiatric disorder that would prevent communication
* volunteered to participate in the study

Exclusion Criteria:

* Patients who were known to present difficulties when entering the fistula (requiring multiple cannulations)
* had a history of hematoma or stenosis in the AVF
* had an infection at the fistula site
* took painkillers within 3 hours of treatment
* did not want to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Invasive pain | Up to two weeks
  It will be assessed three times at the end of the dialysis session with Visual Analogue. Pain intensity measured on a Visual Analog Scale with scores ranging from 0 - 10. Pain increases as the score increases. The high point describes bad outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Ozen, Assoc. Prof., Principal Investigator — Istanbul Demiroglu Bilim University
Locations (1):
- Demiroglu Bilim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozen N, Tosun B, Sayilan AA, Eyileten T, Ozen V, Ecder T, Tosun N. Effect of the arterial needle bevel position on puncture pain and postremoval bleeding time in hemodialysis patients: A self-controlled, single-blind study. Hemodial Int. 2022 Oct;26(4):503-508. doi: 10.1111/hdi.13044. Epub 2022 Sep 6. PMID 36068183
- [Background] Sadeghpour Marvi H, Baloochi Beydokhti T, Sajjadi M, Khaleghimanesh B. Comparing Effects of Rhythmic Breathing and Lidocaine Spray on Pain Intensity During Needle Insertion Into Arteriovenous Fistula in Hemodialysis Patients: A Randomized Controlled Trial. Anesth Pain Med. 2023 Apr 17;13(2):e126384. doi: 10.5812/aapm-126384. eCollection 2023 Apr. PMID 37645007